CLINICAL TRIAL: NCT01103466
Title: A Randomised Controlled Cross-over Study Investigating the Performance and Safety of the Ostomy Base Plate SSH
Brief Title: Investigation of the Performance of Ostomy Base Plate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP204OC
Record Dates: First submitted 2010-04-13; First posted 2010-04-14 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Ileostomy - Stoma
Keywords: Ileostomy base plate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- New ostomy appliance (Atlas) (Active Comparator): Atlas= new base plate. Due to company confidentiality the product is just called Atlas and this is not short for any other names
  Interventions: Device: Atlas
- SenSura (Active Comparator): Commercially available ostomy appliance
  Interventions: Device: SenSura
- Conform 2 (Active Comparator): Commercially available ostomy appliance
  Interventions: Device: Conform 2

INTERVENTIONS:
Device: Atlas — Altas base plates are tested for 14 days (minimum 4 base plates) and the degree of leakage under the baseplate is measured and compared to two other types of base plates.
  Other Names: ostomy appliance
  Arms: New ostomy appliance (Atlas)
Device: SenSura — SenSura base plates are tested for 14 days (minimum 4 base plates) and the degree of leakage under the baseplate is measured and compared to two other types of base plates.
  Other Names: ostomy appliance
  Arms: SenSura
Device: Conform 2 — Conform 2 base plates are tested for 14 days (minimum 4 base plates) and the degree of leakage under the baseplate is measured and compared to two other types of base plates.
  Other Names: Ostomy appliance
  Arms: Conform 2

SUMMARY:
The purpose of this study is to evaluate the performance of Atlas (new base plate) on the degree of leakage under the base plate compared to SenSura and Conform 2. Our hypothesis is that Atlas will do better than the two comparator products.

DETAILED DESCRIPTION:
Peristomal skin problems are reported to have a negative impact on the quality of life of people with a stoma and cause one third of all visits to a stoma care nurse. Stoma effluent in contact with the peristomal skin (leakage) appears to predispose patients to peristomal skin problems. To protect the skin against effluent, the appliance used for collection of stoma effluent should completely cover the peristomal skin close to the stoma. Coloplast has developed a new base plate (SSH) to improve security and increase comfort by minimizing leakage (seeping under the base plate) risk and thereby also the leakage related peristomal skin problems.

The purpose with this clinical study is to evaluate the effect of the new base plate on the degree of leakage under the base plate compared to two existing base plates on the market.

The study is a randomised controlled cross-over intervention study, where all study participants will test all three test products (SSH, Conform 2 and Sensura). Each test period will last 14 days. If 4 changes of base plates is not obtained during the 14 days, the test period will be prolonged until 4 base plate changes is obtained. However, the max test period of one type of product is 21 days. The participants will visit the study investigator at study start and at every shift to a new type of test product. At these visits they will answer questions about the tested product, have a peristomal skin examination and be instructed in how to use the next test products for the next treatment period. Evaluation of leakage and handling will occur via questionnaires the participants take home.

80 healthy participants with an ileostomy will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written Informed Consent
2. Are at least 18 years old
3. Had their ileostomy for minimum 3 months with a size between 20-40 mm
4. Have mental capacity to understand study guidelines and questionnaires
5. Are capable to changing base plate and pouches without help. The help of a caregiver is accepted.
6. Experience leakage under the base plate at least one a week
7. Are currently using a flat 2-piece base plate with mechanical coupling
8. Have been evaluated by investigator (i.e. a health care professional) to have a stoma and peristomal skin condition that is acceptable for entering the study

   -

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Currently suffering from peristomal skin problems where the skin is damaged or bleeding (red and broken / broken and bleeding) as clinically evaluated by the investigator.
3. Currently receiving or have within the past 2 months received radio- and/or chemotherapy
4. Currently using steroid product on peristomal skin (injections and oral treatment are accepted)
5. Currently using a convex system
6. Participating in other clinical studies or have previously participated in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lis H Poulsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Herlev Hospital, Herlev, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a user database in Denmark.
Pre-assignment Details: 41 subjects were enrolled, however 6 subjects did not comply with the inclusion and exclusion criteria. Four of these were terminated before testing any products. Whereas two subjects were included in the safety population as the inclusion criteria violation was first discovered after they tested a product.
Groups:
- Atlas: New base plate
  All subjects tested this test product in one period during the study.
  No parcipitants recieved the same study intervention more than once
- SenSura; Conform2: Commercially available base plate
  All subjects tested this test product in one period during the study.
  No parcipitants recieved the same study intervention more than once
Period: First Period (14 +/- 3 Days)
Arm/Group | Atlas | SenSura | Conform2
Started | 12 | 12 | 13
Completed | 10 | 12 | 13
Not Completed | 2 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Period: Second Period (14 +/- 3 Days)
Arm/Group | Atlas | SenSura | Conform2
Started | 15 | 13 | 7
Completed | 13 | 11 | 6
Not Completed | 2 | 2 | 1
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 1
Period: Third Period (14 +/- 3 Days)
Arm/Group | Atlas | SenSura | Conform2
Started | 8 | 8 | 14
Completed | 6 | 8 | 13
Not Completed | 2 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — not satisfied with product | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 2 subjects were excluded from the ITT and PP population, and therefore not included in the baseline measurements
Groups:
- All Study Parcipitants: All parcipitants recieved all three intervention and they are therefore combined into one group.
Arm/Group | All Study Parcipitants
Number analyzed (Participants) | 35
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Leakage Under the Base Plate
Description: Area of leakage under the base plate is recorded on a circular scale going from 0 fields to 24 fields where 0 is "no leakage" and 24 is "complete leakage" under the base plate.
Time Frame: At every change of base plate
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Atlas: new base plate
- SenSura; Conform2: base plate
Arm/Group | Atlas | SenSura | Conform2
Number analyzed (Participants) | 35 | 33 | 34
units on a scale | 8.2 (5.0) | 5.5 (4.8) | 8.0 (4.9)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from inclusion to the end of the three test periods (~43 days).
Description: The safety population contained 37 subjects, whereof two subjects were excluded from the ITT population due to inclusion criteria violation and did not try any test products.
Arm/Group | Atlas | SenSura | Conform2
Serious Adverse Events (participants affected / at risk) | 2/35 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 6/35 | 1/33 | 6/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atlas (N=35) | SenSura (N=33) | Conform2 (N=34)
Volvulus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atlas (N=35) | SenSura (N=33) | Conform2 (N=34)
skin irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 6 (7)
faeces leakage under base plate (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes